CLINICAL TRIAL: NCT06596473
Title: A Multicenter, Open-Label, Phase 1a/b First-in-Human Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BG-C477 in Patients With Selected Advanced Solid Tumors
Brief Title: A Study of BG-C477 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-C477-101; CTR20244563 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
Keywords: BG-C477; advanced solid tumors; CEA ADC
MeSH Terms: interventions — tislelizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a: BG-C477 Monotherapy Dose Escalation (Experimental): Sequential cohorts of increasing dose levels of BG-C477 will be evaluated as monotherapy.
  Interventions: Drug: BG-C477
- Phase 1a: BG-C477 Monotherapy Safety Expansion (Experimental): Selected dose levels that have been determined to be safe in Phase 1a dose escalation will be further evaluated in monotherapy.
  Interventions: Drug: BG-C477
- Phase 1b Part A: BG-C477 Monotherapy Expansion and Dose Optimization (Experimental): Participants with selected advanced solid tumors will be evaluated at different dose levels of RDFEs identified in Phase 1a.
  Interventions: Drug: BG-C477
- Phase 1b Part B: Combination Therapy Expansion (Experimental): Sequential cohorts of increasing dose levels of BG-C477 will be evaluated in combination with anticancer agents, including chemotherapy or tislelizumab.
  Interventions: Drug: BG-C477; Drug: Tislelizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: BG-C477 — Administered intravenously.
Drug: Tislelizumab — Administered intravenously.
  Other Names: BGB-A317
  Arms: Phase 1b Part B: Combination Therapy Expansion
Drug: Chemotherapy — Administered in accordance with relevant local guidelines and/or prescribing information.
  Arms: Phase 1b Part B: Combination Therapy Expansion

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of BG-C477 alone and in combination with anticancer agents in participants with selected advanced solid tumors.

DETAILED DESCRIPTION:
This new study will check how safe and helpful a potential anticancer drug called BG-C477 is. This drug will be tested by itself or combined with other anticancer agents. The purpose of this study is to test if BG-C477 is safe and if it works in people with your disease when it is given on its own and in combination with other anticancer agents.

Note: Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign the informed consent form (ICF) and be capable of giving written informed consent
* Participants must consent to provide an archival tumor tissue sample or a fresh baseline biopsy
* Phase 1a (Dose Escalation): Histologically confirmed advanced, metastatic, or unresectable solid tumors, that were previously treated with at least 2 lines of standard systemic therapy or for whom no standard treatment is available in the medical judgment of the investigator
* Phase 1b (Dose Expansion) Part A: Histologically confirmed advanced or metastatic select solid tumors that were previously treated with and progressed from at least 1 line of standard systemic therapy
* Phase 1b (Dose Expansion) Part B: Histologically confirmed advanced or metastatic select solid tumors who have previously received 0 or 1 line of systemic therapy for advanced disease
* ≥ 1 measurable lesion as assessed by RECIST v1.1
* Stable Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Adequate organ function
* Female participants of childbearing potential must be willing to use a highly effective method of birth control and refrain from egg donation for the duration of the study and for ≥ 8 months after the last dose of BG-C477, for ≥ 6 months after the last dose of chemotherapy, and for ≥ 4 months after the last dose of tislelizumab,whichever comes later
* Nonsterile male participants must be willing to use a highly effective method of birth control and refrain from sperm donation for the duration of the study and for ≥ 5 months after the last dose of BG-C477, for ≥ 3 months after chemotherapy, and for ≥ 4 months after the last dose of tislelizumab, whichever comes later.

Exclusion Criteria:

* Prior treatment with any carcinoembryonic antigen (CEA)-targeted ADCs or ADCs containing topoisomerase 1 (TOP1) inhibitor as payload
* History of severe allergic reactions, severe reaction to infusion, or hypersensitivity to the active ingredient and excipients of the study drug(s) or protein-based therapeutics
* Active leptomeningeal disease or uncontrolled, untreated brain metastasis
* Any malignancy ≤ 2 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose of the study drug(s) to 30 days after the last dose (up to approximately 2 years)
  Number of participants with AEs and SAEs, including findings from abnormal laboratory assessments, and that meet protocol-defined dose-limiting toxicity (DLT) criteria or protocol-defined Adverse Event of Clinical Interest (AECI) criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) | Approximately 1 year
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended Dose(s) for Expansion (RDFE[s]) of BG-C477 | Approximately 1 year
  RDFE of BG-C477 monotherapy will be determined based upon available data.
Phase 1b: Overall Response Rate (ORR) | Approximately 2 years
  ORR is defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR), as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Phase 1b: Recommended Phase 2 Dose (RP2D) of BG-C477 | Approximately 2 years
  RP2D of BG-C477 alone and in combination with anticancer agents will be determined based upon available data.

SECONDARY OUTCOMES:
Phase 1a: ORR | Approximately 1 year
  ORR is defined as the percentage of participants with best overall response of CR or PR, as assessed by the investigator per RECIST v1.1.
Phase 1a and 1b: Duration of Response (DOR) | Approximately 2 years
  DOR is defined as the time from the first determination of an objective response until first documentation of disease progression or death due to any cause, whichever occurs first, as assessed by the investigator per RECIST Version 1.1.
Phase 1a and 1b: Disease Control Rate (DCR) | Approximately 2 years
  DCR is defined as the percentage of participants who achieve best overall response of CR, PR, or stable disease, as assessed by the investigator per RECIST Version 1.1.
Phase 1b: Progression-Free Survival (PFS) | Approximately 2 years
  PFS is defined as the time from the first administration of study drug(s) to the date of first documentation of disease progression or death due to any cause, whichever occurs first, as assessed by the investigator per RECIST Version 1.1.
Phase 1b: Number of Participants with AEs and SAEs | From first dose of the study drug(s) to 30 days after the last dose (up to approximately 2 years)
  Number of participants with AEs and SAEs, including findings from physical examinations, laboratory assessments, and that meet protocol-defined DLT criteria or protocol-defined AECI criteria.
Phase 1a and 1b: Maximum observed plasma concentration (Cmax) of BG-C477 antibody-drug conjugate (ADC), BG-C477 total antibody, and free payload | Approximately 2 months
Phase 1a and 1b: Minimum concentration (Cmin) of BG-C477 | Approximately 2 months
Phase 1a and 1b: Time to reach maximum observed plasma concentration (Tmax) of BG-C477 | Approximately 2 months
Phase 1a and 1b: Area under the concentration-versus-time curve during dosing interval (AUCtau) of BG-C477 | Approximately 2 months
Phase 1a and 1b: Apparent terminal elimination half-life (t1/2) of BG-C477 | Approximately 2 months
Phase 1a and 1b: Systemic clearance (CL/F) of BG-C477 | Approximately 2 months
Phase 1a and 1b: Apparent volume of distribution at steady state (Vss) of BG-C477 | Approximately 2 months
Phase 1a and 1b: Number of Participants with Antidrug Antibodies (ADAs) against BG-C477 | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (16):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - The University of Kansas Cancer Center, Westwood, Kansas
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Cancer Research South Australia, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - One Clinical Research, Nedlands, Western Australia
- China (7):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical Universitywuxiang Branch, Nanning, Guangxi
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - Jining No Peoples Hospital East Branch, Jining, Shandong
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/